CLINICAL TRIAL: NCT03250169
Title: Neurofilament Heavy and Light Chain Testing for NEDA (No Evidence of Disease Activity) Assessing in Multiple Sclerosis: a Longitudinal Biomarker Study
Brief Title: Neurofilaments for NEDA Assessing in MS
Status: Terminated | Type: Observational
Why Stopped: Under recruitment
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 011717
Record Dates: First submitted 2017-07-19; First posted 2017-08-15 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alemtuzumab — Licensed dose

SUMMARY:
Goal is to evaluate the achievement of biological NEDA as demonstrated by a drop in neurofilament levels in MS patients commencing Alemtuzumab therapy as part of their MS management.

DETAILED DESCRIPTION:
Primary

1. To evaluate the achievement of NEDA using blood and CSF neurofilaments in Alemtuzumab treated patients.

   Secondary
2. To assess prognosis at the end of the study based on neurofilament status.
3. To correlate neurofilament levels with clinical and MRI markers of disease activity.
4. To evaluate the effect of Alemtuzumab on the profile of other CSF, blood, urine, faeces biomarkers of inflammation, neurodegeneration, neuronal sprouting and synaptogenesis, treatment activity and metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Relapsing Remitting Multiple Sclerosis (RRMS).
2. Age 18-55 years.
3. EDSS score between 0-5.5.
4. Commencing Alemtuzumab therapy at Neurology Infusion and Planned Investigation Unit, The Royal London Hospital, Ward 11D

Exclusion Criteria:

1. A diagnosis of Secondary Progressive MS (SPMS) or other forms of progressive MS.
2. Those unable to comply with study requirement

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Relapsing-remitting MS
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Blood and CSF neurofilaments in Alemtuzumab patients over 24months | 2 years
  Neurofilaments

SECONDARY OUTCOMES:
Overall clinical response based on neurofilament response | 2 years
  neurofilaments
Neurofilament status and association with clinical and MRI markers of disease activity. | 2 years
  Correlation index
Longitudinal assessment of other biomarkers of inflammation & plasticity | 2 years
  Correlation index

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No